CLINICAL TRIAL: NCT04672603
Title: Effects of Complete Preservation Versus Partial Preservation of Denonvilliers' Fascia on Postoperative Urogenital Function in Locally Advanced Non-anterior Mid-low Rectal Cancer Patients：A Multicenter，Randomized Study
Brief Title: Complete Versus Partial Preservation of Denonvilliers' Fascia on Urogenital Function in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UGFS-01
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer; Advanced Cancer
Keywords: Urogenital Function; Denonvilliers' Fascia
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Preservation of Denonvilliers Fascia (Experimental): Complete preservation of Denonvilliers fascia in Laparoscopy-assisted pelvic autonomic nerve preservation surgery with TME for mid-low rectal cancer patients.
  Interventions: Procedure: Complete Preservation of Denonvilliers' Fascia
- Partial Preservation of Denonvilliers Fascia (No Intervention): Partial preservation of Denonvilliers fascia in Laparoscopy-assisted pelvic autonomic nerve preservation surgery with TME for mid-low rectal cancer patients.

INTERVENTIONS:
Procedure: Complete Preservation of Denonvilliers' Fascia — Patients accept L-PANP surgery with complete preservation of Denonvilliers Fascia
  Arms: Complete Preservation of Denonvilliers Fascia

SUMMARY:
Total mesorectal resection (TME) is the standard surgical method for locally advanced rectal cancer, which significantly reduces the local recurrence rate. However, the incidence of urogenital dysfunction is higher. Studies found that Denonvilliers' Fascia contains autonomic nerves that may regulate urogenital function, while traditional TME surgery resects part of it. Recent Studies found that complete preservation of Denonvilliers' Fascia could improve urogenital in selected patients with rectal cancer. Locally advanced patient (T3-4 and/or N+, M0) accounts for a high proportion of mid-low rectal cancer. However, whether these patients can benefit from it has not fully been demonstrated. This project conducts a multi-center randomized controlled study to evaluate the effects of complete preservation and partial preservation of Denonvilliers' Fascia on postoperative urogenital function of locally advanced non-anterior mid-low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of rectal adenocarcinoma;
2. Preoperative staging cT3-4 and or N+，M0 rectal cancer (AJCC- 7th);
3. Non-anterior wall, mid-low rectal cancer from 0 to 12 cm from the anal verge measured by rigid proctoscope;
4. R0 surgical results is expected by transabdominal or transanal TME/TSME;
5. 18 < age (years) < 71, informed consent;
6. Normal erection function (IIEF-5>21), ejaculation function grading as I level, FSFI > 26, normal urinary function (Bladder residual urine<100ml);
7. Preoperative ASA grade I ~ III, no serious systemic disease;

Exclusion Criteria:

1. Preoperatively confirmed peritoneum or distant metastasis;
2. Intraoperative confirmed invasion of surrounding tissues or organs, cannot be R0 resected;
3. With other malignant diseases;
4. With acute ileus, perforation or hemorrhage,need emergency surgery;
5. Critical organs dysfunction, unable to tolerate laparoscopic surgery;
6. With severe mental illness, cannot be evaluated;

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of sexual dysfunction | 1 month
  IIEF-5(International questionnaire of erectile function-5), Ejaculation function and FSFI questionnaires are used to assess sexual function
Incidence of urinary dysfunction | 1 month
  IPSS(International prostate symptom score), ICIQ, bladder residual urine volume and urodynamic study are used to assess urinary function

SECONDARY OUTCOMES:
Incidence of sexual dysfunction | 9 months
  IIEF-5, Ejaculation function and FSFI questionnaires are used to assess sexual function
Incidence of urinary dysfunction | 9 months
  IPSS, ICIQ questionnaires, bladder residual urine volume and urodynamic study are used to assess urinary function
Quality of life assessed with GIQLI questionnaires | 1month
  GIQLI questionnaires are used to assess quality of life
Quality of life assessed with GIQLI questionnaires | 9 months
  GIQLI questionnaires are used to assess quality of life
1-year local recurrence | 1 year
  1-year local recurrence
1-year overall survival rate | 1 year
  1-year overall survival rate
Positive Circumferential Resection Margin Rate | 1 week
  Positive Circumferential Resection Margin Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China